CLINICAL TRIAL: NCT03002740
Title: Bleeding Events and Oral Anticoagulant Treatment in Non-Valvular Atrial Fibrillation (Heart-BEAT): A Cohort Study Based on CPRD-HES Data
Brief Title: Bleeding Events and Oral Anticoagulant Treatment in Non-Valvular Atrial Fibrillation
Status: Withdrawn | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-491
Record Dates: First submitted 2016-12-21; First posted 2016-12-26 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Non-valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- NVAF patients newly prescribed apixaban
- NVAF patients newly prescribed rivaroxaban
- NVAF patients newly prescribed dabigatran
- NVAF patients newly prescribed VKA

SUMMARY:
In a population of patients with non-valvular atrial fibrillation (NVAF), and treated with oral anticoagulants (OAC) in routine clinical practice in England, this study will describe patients treated with each OAC, and to estimate and compare event rates of treatment discontinuation, bleeding, and healthcare resource utilisation (HCRU) across OAC treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Have a prescription for apixaban, rivaroxaban, dabigatran, or VKA during the study period
2. Are ≥ 18 years of age at index date
3. Have ≥ 12 months of computerised medical data prior to index date (date of OAC initiation)
4. Have a record of AF on or ever prior to index date

Exclusion Criteria:

1. Have a record for a valvular condition that is considered causal for AF on or ever prior to index date
2. Have a history of the OACs which are prescribed during the study period (ie, history of index OAC, as patients need to be newly prescribed either apixaban, rivaroxaban, dabigatran, or VKA)
3. Have more than 1 OAC exposure which starts on the same date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with NVAF recorded in the UK Clinical Practice Research Datalink(CPRD) and Hospital Episode Statistics(HES) database, and who were newly prescribed with apixaban, rivaroxaban, dabigatran or VKA from 1st December 2012 and 31st December 2015 (or up to the most recent data available).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of clinically relevant bleeding events following treatment initiation among NVAF patients newly prescribed oral anticoagulants (OACs) | Approximately 3 years

SECONDARY OUTCOMES:
Composite of clinical characteristics in patients with non-valvular atrial fibrillation (NVAF) newly prescribed oral anticoagulants (OACs) | At baseline
Composite of patient demographics in patients with non-valvular atrial fibrillation (NVAF) newly prescribed oral anticoagulants (OACs) | At baseline
Cumulative incidence of a major bleeding event following treatment initiation among NVAF patients newly prescribed oral anticoagulants (OACs) | Approximately 3 years
Cumulative incidence of a thromboembolic event following treatment initiation among NVAF patients newly prescribed oral anticoagulants (OACs) | Approximately 3 years
Composite of Healthcare resource utilization patients newly prescribed oral anticoagulants (OACs) | Approximately 3 years
  Healthcare resource utilization corresponds to referrals, hospitalizations, prescriptions, and laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx